CLINICAL TRIAL: NCT03111030
Title: ProACTIVE SCI Physical Activity Coaching Intervention
Brief Title: ProACTIVE SCI Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Rick Hansen Institute (Other); Ontario Neurotrauma Foundation (Other); International Collaboration on Repair Discoveries (Other)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-00559
Record Dates: First submitted 2017-03-16; First posted 2017-04-12 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProacTive SCI (Experimental): Individualized physical activity coaching sessions
  Interventions: Behavioral: ProacTive SCI
- Wait-list control (No Intervention): Standard care, receiving physical activity coaching sessions after completing post-testing

INTERVENTIONS:
Behavioral: ProacTive SCI — Participants will receive weekly physical activity coaching sessions. Each session will be 10-15 minutes, delivered either face to face, over Skype, or over the phone. Additional resources may be emailed to participants based on need throughout the intervention (for example, a goal, list of places to exercise, contact information to reach mentoring services). A typical session may include:
  1. An assessment of motivated the participant is to be physically active
  2. A: If motivated, a physical activity goal will be set, strategies will be reviewed, and resources to accomplish that goal will be provided.
     B: If not motivated, questions will be asked to understand why the reasons for lack of motivation. If it is for any reasons including barriers, fear, confidence, or knowledge, the interventionist will discuss strategies to overcome these obstacles.
  3. Progress and barriers will be reassessed and discussed.
  Arms: ProacTive SCI

SUMMARY:
This study will employ a randomized, wait-list controlled trial. A total of 30 participants (15 experimental, 15 wait-list control) between 18-65 years of age who have chronic SCI ≥ 1 year prior will be recruited. Physical activity measures will be taken using wrist-based accelerometers and the Leisure Time Physical Activity Questionnaire for people with SCI (LTPAQ). Psychosocial factors will be evaluated through questionnaires. The primary health outcome measure (aPWV), and secondary cardiovascular parameters will be assessed using a combination of echocardiography and ultrasound. Fitness will be determined using a peak oxygen consumption test on an arm-cycle ergometer. All measurement will be taken at baseline and after 9 weeks following intervention commencement. Physical activity will also be sampled mid-intervention at 4 and 7 weeks. Training will involve weekly, 10-15 minute coaching sessions for 9 weeks. All pre- and post-assessments will take place at the Blusson Spinal Cord Centre at ICORD. Intervention content will be delivered in-person, over Skype or phone, and the wrist- worn accelerometers will be delivered and picked up from the participant's home during the intervention.

DETAILED DESCRIPTION:
A randomized, wait-list controlled trial will be used to compare the effects of tailored PA coaching sessions versus no coaching on PA behaviour, psychosocial factors, and health outcomes. Eligible individuals will be randomly assigned (1:1) to either the experimental (PA coaching sessions) or wait-list control condition. Matched randomization based on baseline physical activity levels will be used. The randomization sequence will be generated by a research assistant independent of the trial.

Day 1 testing measures include vascular measures (arterial pulse wave velocity, arterial structure; 30 minutes), cardiac structure and function measures (30 minutes), a peak oxygen uptake test (60 minutes), for a total duration of 2 hours. Participants will be given an accelerometer to wear for the 6-day monitoring period (6.1.2) after which they will return for Day 2 testing.

Day 2 testing measures include administration of the LTPAQ (5 minutes), administration of the demographics and Health Action Process Approach model questionnaire (25 minutes), and a measurement of energy expenditure at different sub-maximal wheeling speeds to calibrate MVPA cut-points (30 minutes) and at baseline, the first PA coaching session will be administered (60 minutes) whereas at post-test a semi-structured interview will be administered (60 minutes). Total duration of day 2 testing will be 2 hours. The intervention protocol is described below. During the intervention, physical activity will be sampled at two time points; accelerometer and PARA SCI data will be taken during week 4 and week 7.

INTERVENTION

Intervention Protocol:

Experimental participants will receive weekly PA coaching sessions. Each session will be 10-15 minutes in duration and delivered either face to face, over Skype, or when the former modes are unavailable, over the phone. Additionally, supplemental resources may be emailed to the participants based on need throughout the intervention.

Participants' motivation to exercise will first be determined according to stages of the HAPA model. Those who identify as pre-intenders (no intention to exercise) will receive intervention strategies that focus on changing motivation to be physically active. Those identified as intenders (willing to exercise but have not started) will focus on providing resources and behavioural strategies to commence physical activity. Lastly, those identified as actors (already exercising) will receive intervention strategies that help participants maintain or improve PA behaviour.

For those in the intender or actor stage, the intervention aims to promote the international SCI PA guidelines to promote fitness (at least 20 minutes of moderate vigorous aerobic activity twice/week and strength training twice/week). For those exceeding the fitness guidelines, the international SCI PA guidelines to promote health are promoted (at least 30 minutes of moderate to vigorous aerobic activity three times/week and strength training twice/week). However, these aims will be modified based on the individual's baseline PA. During the first visit, participants' baseline PA levels will be reviewed and an appropriate PA goal to achieve in the following month will be formed. Ultimately, the goal is the decision of the participant.

Following goal setting, barriers to participating in PA will be identified. The interventionist will select intervention strategies based on the identified barriers. A pre-formed chart of corresponding intervention strategies (e.g. use of behaviour change techniques, referral to facilities or peers, suggesting at-home exercises) was developed to aid this pairing process (Appendix A). These intervention strategies are accompanied by a comprehensive toolkit based from the HAPA model (Appendix B). In brief, the toolkit advises on three key strategies for promoting PA to people with SCI: i) education, ii) referral, iii) tailored PA prescription.

Remaining weekly coaching sessions will review participants' progress and barriers to discuss new goals and strategies as outlined above.

Control Participants:

Control participants will complete baseline and post-testing only. Following completion of post-test measures they will be administered the same PA coaching session as the intervention group, with post-test measures being repeated upon intervention completion.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be competent to give informed consent,
* be able to propel an arm ergometer.

Exclusion Criteria:

* History and/or symptoms of CVD or cardiopulmonary problems/disease.
* Major trauma or surgery within the last 6 months.
* Active Stage 3 or 4 pressure ulcer (based on the National Pressure Ulcer Advisory Panel classification)
* Recent (within 1 year) history of lower-extremity or non-union fracture
* Any unstable medical/psychiatric condition or substance abuse disorder that is likely to affect their ability to complete this study.
* Individuals with active medical issues such as pressure sores, urinary tract infections, hypertension, or heart disorders.
* Any cognitive dysfunction or language barrier that would prevent subjects from following English instructions.
* Subjects may be excluded at the discretion of the principal investigator due to other, unforeseen, safety issues.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants may self- identify as male, female, other
Enrollment: 28 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Martin Ginis, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (2):
- Canada (2):
  - University of British Columbia Okanagan, Kelowna, British Columbia
  - International Collaboration on Repair Discoveries, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoekstra F, Martin Ginis KA, Collins D, Dinwoodie M, Ma JK, Gaudet S, Rakiecki D; SCI Exercise Counselling Panel; Gainforth HL. Applying state space grids methods to characterize counsellor-client interactions in a physical activity behavioural intervention for adults with disabilities. Psychol Sport Exerc. 2023 Mar;65:102350. doi: 10.1016/j.psychsport.2022.102350. Epub 2022 Dec 9. PMID 37665832
- [Derived] Dinwoodie M, Hoekstra F, Stelzer S, Ma JK, Martin Ginis KA. A dynamic analysis of physical activity barriers experienced by adults with spinal cord injury. Spinal Cord Ser Cases. 2022 Mar 29;8(1):37. doi: 10.1038/s41394-022-00504-y. PMID 35351871
- [Derived] Hoekstra F, Collins D, Dinwoodie M, Ma JK, Martin Ginis KA. Measuring behavior change technique delivery and receipt in physical activity behavioral interventions. Rehabil Psychol. 2022 May;67(2):128-138. doi: 10.1037/rep0000440. Epub 2022 Mar 17. PMID 35298203
- [Derived] Ma JK, West CR, Martin Ginis KA. The Effects of a Patient and Provider Co-Developed, Behavioral Physical Activity Intervention on Physical Activity, Psychosocial Predictors, and Fitness in Individuals with Spinal Cord Injury: A Randomized Controlled Trial. Sports Med. 2019 Jul;49(7):1117-1131. doi: 10.1007/s40279-019-01118-5. PMID 31119717

RESULTS

PARTICIPANT FLOW:
Groups:
- ProacTive SCI: Individualized physical activity coaching sessions
  ProacTive SCI: Participants will receive weekly physical activity coaching sessions. Each session will be 10-15 minutes, delivered either face to face, over Skype, or over the phone. Additional resources may be emailed to participants based on need throughout the intervention (for example, a goal, list of places to exercise, contact information to reach mentoring services). A typical session may include:
  1. An assessment of motivated the participant is to be physically active
  2. A: If motivated, a physical activity goal will be set, strategies will be reviewed, and resources to accomplish that goal will be provided.
     B: If not motivated, questions will be asked to understand why the reasons for lack of motivation. If it is for any reasons including barriers, fear, confidence, or knowledge, the interventionist will discuss strategies to overcome these obstacles.
  3. Progress and barriers will be reassessed and discussed.
Period: Overall Study
Arm/Group | ProacTive SCI | Wait-list Control
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProacTive SCI | Wait-list Control | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.79 (13.63) | 45.57 (10.49) | 45.68 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 0 | 0 | 0
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 14 | 28
Leisure Time Physical Activity Questionnaire for People With SCI (LTPAQ) [Mean (Standard Deviation); unit: Total LTPA min/week] — Participants will be asked to complete a questionnaire, guided by the co-investigator (Jasmin Ma), that asks the participant to recall in the last 7 days how many days and for how long leisure time physical activity was performed. The recall assessment will take approximately 5 minutes to complete.
  Total LTPA min/week | 212 (195) | 274 (300) | 243 (248)
Aerobic Fitness Evaluation: Peak Oxygen Uptake Test (VO2peak) [Mean (Standard Deviation); unit: L/min] | 1.15 (.36) | 1.13 (.43) | 1.14 (.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity: Leisure Time Physical Activity Questionnaire for People With SCI (LTPAQ)
Description: Participants will be asked to complete a questionnaire, guided by the co-investigator (Jasmin Ma), that asks the participant to recall in the last 7 days how many days and for how long leisure time physical activity was performed. The recall assessment will take approximately 5 minutes to complete.
Time Frame: Baseline, week 4, week 7, week 10, 6 month follow up
Measure: Mean (Standard Deviation); unit: Total LTPA min/week
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
Total LTPA min/week
  Baseline | 212 (195) | 274 (300)
  Week 4 | 393 (413) | NA (NA) — Data only collected in intervention group
  Week 7 | 370 (258) | NA (NA) — Data only collected in intervention group
  Week 10 | 405 (364) | 147 (192)
  6 months FU | 348 (269) | NA (NA) — Data only collected in intervention group

2. Primary Outcome: Change in Total Accelerometer Count as a Measure of Change in Physical Activity: 6-day Physical Activity Monitoring Period
Description: Participants will be fitted with a wrist-based tri-axial accelerometer to be worn 24 hours a day for 6 days in order to determine intensity and amount of PA. They will keep a detailed PA diary recording all leisure time PA performed during the day. The primary outcome will be total vector magnitude (VM) accelerometer counts from a tri-axial wrist-worn accelerometer (GT9X, ActiGraph LLC, FL). During the intervention, the accelerometer will be picked up and dropped off to the participant's home to decrease burden. Text or email reminders (i.e. "Please don't forget to wear your accelerometer today") will be used to promote adherence to accelerometer wear.
Time Frame: Baseline, week 4, week 7, week 10
Measure: Mean (Standard Deviation); unit: Accelerometer total VM counts
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
Accelerometer total VM counts
  Baseline | 562000 (188000) | 848000 (759000)
  Week 4 | 593000 (307000) | NA (NA) — Data only collected in intervention group
  Week 7 | 659000 (338000) | NA (NA) — Data only collected in intervention group
  Week 10 | 702000 (267000) | 598000 (390000)

3. Secondary Outcome: Change in Health Action Process Approach Model Measure
Description: This survey will examine psychological factors that may affect PA participation. The survey will be recorded either electronically or with pen and paper depending on the respondent's preference. Survey will take approximately 25 minutes to complete, and will assess constructs related to exercise such as perceived risks, self- efficacy, planning, and social support. The demographics questionnaire will also be administered with this measure. All items will be assessed on a 7-point Likert scale ranging from 1 = "strongly disagree" to 7 = "strongly agree". Higher scores indicate a better outcome.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Affective outcome expectancies (Baseline) | 5.1 (1.3) | 5.7 (0.9)
  Affective outcome expectancies (Week 10) | 5.6 (1.0) | 5.4 (1.0)
  Instrumental outcome expectancies (Baseline) | 6.5 (0.6) | 6.5 (0.9)
  Instrumental outcome expectancies (Week 10) | 6.8 (0.3) | 6.3 (0.8)
  Risk perceptions (Baseline) | 2.5 (1.6) | 2.5 (1.3)
  Risk perceptions (Week 10) | 2.8 (1.6) | 2.5 (1.1)
  Aerobic exercise task self-efficacy (Baseline) | 3.4 (1.9) | 4.1 (1.7)
  Aerobic exercise task self-efficacy (Week 10) | 4.7 (1.2) | 3.6 (1.6)
  Strength exercise task self-efficacy (Baseline) | 3.9 (1.6) | 3.7 (1.6)
  Strength exercise task self-efficacy (Week 10) | 5.6 (1.2) | 3.2 (1.8)
  Intentions (Baseline) | 6.1 (1.1) | 6.5 (0.7)
  Intentions (Week 10) | 6.8 (0.4) | 6.3 (1.2)
  Planning self-efficacy (Baseline) | 5.9 (0.8) | 6.2 (1.1)
  Planning self-efficacy (Week 10) | 6.0 (0.5) | 6.8 (0.4)
  Barrier self-efficacy (Baseline) | 5.0 (1.2) | 4.4 (1.0)
  Barrier self-efficacy (Week 10) | 5.7 (0.8) | 4.7 (1.1)
  Scheduling self-efficacy (Baseline) | 4.9 (1.5) | 5.3 (1.2)
  Scheduling self-efficacy (Week 10) | 5.7 (1.3) | 5.5 (1.1)
  Action planning (Baseline) | 3.7 (1.9) | 3.8 (2.0)
  Action planning (Week 10) | 6.8 (0.4) | 3.6 (2.3)
  Monitoring (Baseline) | 4.5 (1.6) | 4.4 (1.4)
  Monitoring (Week 10) | 6.3 (0.8) | 4.4 (1.3)
  Coping self-efficacy (Baseline) | 6.0 (0.8) | 5.8 (1.2)
  Coping self-efficacy (Week 10) | 6.3 (0.7) | 6.3 (0.7)
  Social support (Baseline) | 2.2 (1.0) | 2.0 (0.8)
  Social support (Week 10) | 2.8 (0.9) | 1.7 (0.5)
  Presence of barriers (Baseline) | 5.7 (1.5) | 5.5 (1.3)
  Presence of barriers (Week 10) | 6.1 (1.1) | 5.0 (1.8)
  Knowledge (Baseline) | 5.9 (1.1) | 5.2 (1.9)
  Knowledge (Week 10) | 6.7 (0.4) | 4.4 (2.0)

4. Secondary Outcome: Number of Participants Participating in Qualitative Interviews
Description: A semi-structured interview will be conducted at the end of the intervention to understand what components were and were not effective. Data will not be recorded. This feedback will be used to improve future iterations of the intervention. There is no associated scale with this measurement.
Time Frame: 9 weeks from intervention start (week 10)
Measure: Count of Participants; unit: Participants
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
Participants | 14 | 0

5. Secondary Outcome: Change in Pulse Wave Velocity
Description: aPWV (cm/s) is calculated by dividing the distance between measurement sites, by the pulse transit time. Distance between the carotid and femoral arteries will be measured using measuring tape along the surface of the body, held parallel to the testing table. The pulse transit is determined from the arterial blood pressure waves, which are collected at each arterial site. A pen-like device (model SPT-301; Millar Instruments Inc., Houston, TX) will be applied to the carotid and femoral arterial sites using a light pressure to obtain arterial pressure waves. Heart rate will be recorded using a single-lead (lead I) electrocardiogram (ECG) (model ML 123, ADInstruments Inc., Colorado Springs, CO).
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
cm/s
  Baseline | 10.6 (2.9) | 8.0 (2.0)
  Week 10 | 9.7 (2.5) | 8.2 (1.9)

6. Secondary Outcome: Change in Arterial Structure: Wall Thickness
Description: Common carotid arterial images will be collected using B-mode ultrasound (INFO) for 10 cardiac cycles. Images will be analyzed using internal ultrasound software to determine lumen diameter and intima-media thickness.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
mm
  Baseline | 0.62 (0.16) | 0.56 (0.07)
  Week 10 | 0.61 (0.15) | 0.56 (0.07)

7. Secondary Outcome: Change in End Systolic Volume
Description: Cardiac image will be collected non-invasively using Doppler ultrasound (Vivid q, GE Healthcare, Buckinghamshire, UK). Image will be collected and stored on the ultrasound for offline analysis.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
ml
  Baseline | 38 (9) | 36 (9)
  Week 10 | 38 (9) | 35 (8)

8. Secondary Outcome: Change in End Diastolic Volume
Description: as for outcome 7
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
ml
  Baseline | 87 (18) | 84 (20)
  Week 10 | 86 (14) | 82 (18)

9. Secondary Outcome: Change in Intraventricular Septum Diameter
Description: as for outcome 7
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Population: This was not measured or reported.
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Ventricular Internal Diameter
Description: as for outcome 7
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
mm
  Baseline | 42 (5) | 43 (10)
  Week 10 | 43 (4) | 44 (4)

11. Secondary Outcome: Change in Systolic Function
Description: Cardiac image will be collected non-invasively using Doppler ultrasound (Vivid q, GE Healthcare, Buckinghamshire, UK). Image will be collected and stored on the ultrasound for offline analysis. LV stroke volume will be used to measure change in systolic function.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
ml
  Baseline | 49 (9) | 48 (11)
  Week 10 | 49 (6) | 47 (10)

12. Secondary Outcome: Change in Ejection Fraction
Description: as for outcome 7
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: % of blood ejected per contraction
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
% of blood ejected per contraction
  Baseline | 57 (3) | 57 (3)
  Week 10 | 56 (3) | 58 (3)

13. Secondary Outcome: Change in Cardiac Output
Description: as for outcome 7
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
L/min
  Baseline | 3.22 (0.78) | 3.05 (0.87)
  Week 10 | 3.13 (0.63) | 3.13 (0.96)

14. Secondary Outcome: Change in Fractional Shortening
Description: Cardiac image will be collected non-invasively using Doppler ultrasound (Vivid q, GE Healthcare, Buckinghamshire, UK). Image will be collected and stored on the ultrasound for offline analysis. Longitudinal strain will be used to measure change in fractional shortening.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: % change from original length
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
% change from original length
  Baseline | -19.0 (2.6) | -17.5 (4.3)
  Week 10 | -19.2 (2.7) | -18.1 (3.3)

15. Secondary Outcome: Change in Diastolic Function
Description: Cardiac image will be collected non-invasively using Doppler ultrasound (Vivid q, GE Healthcare, Buckinghamshire, UK). Image will be collected and stored on the ultrasound for offline analysis. E'/A' (ratio between early diastolic septal tissue velocity and late diastolic septal tissue velocity) will be used to measure change in diastolic function.
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
Ratio
  Baseline | 0.99 (0.21) | 1.10 (0.33)
  Week 10 | 1.02 (0.32) | 1.14 (0.36)

16. Secondary Outcome: Aerobic Fitness Evaluation: Peak Oxygen Uptake Test (VO2peak)
Description: Participants will perform a graded arm ergometer test on an electronically braked arm ergometer. For participants with tetraplegia who have limited handgrip function, gloves will be used to secure hands to the ergometer handles. Participants will be instructed to maintain a cycling rate of 50 revolutions per minute (rpm) for the duration of the test. After an initial warm-up at 0W, power output will be increased each minute at a rate of 2-5 W/min for participants with tetraplegia, or 10 W/min for participants with paraplegia, until volitional exhaustion (i.e. dropping below 30 rpm). Oxygen consumption will be recorded on a breath-by-breath basis for the duration of the test and reported as rolling 30-second averages sampled at 5-second intervals as per consensus recommendations.
  All outcome data are reported here: https://doi.org/10.1007/s40279-019-01118-5
Time Frame: Baseline, 9 weeks from intervention start (week 10)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | ProacTive SCI | Wait-list Control
Number analyzed (Participants) | 14 | 14
L/min
  Baseline | 1.16 (0.38) | 1.13 (0.46)
  Week 10 | 1.30 (0.43) | 1.06 (0.40)

ADVERSE EVENTS:
Time Frame: Study duration: 10 weeks
Arm/Group | ProacTive SCI | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03111030/Prot_SAP_000.pdf